CLINICAL TRIAL: NCT05255055
Title: Effectiveness of Therapeutic Exercise Versus Manual Therapy in Patients With Chronic Neck Pain - Randomized Clinical Trial
Brief Title: Effectiveness of Therapeutic Exercise Versus Manual Therapy in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alexander Achalandabaso, Clinical Professor, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAH/2022/01
Record Dates: First submitted 2022-01-20; First posted 2022-02-24 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Chronic Neck Pain
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy Group (Experimental): Manipulation of the high dorsal region in extension. Cervical mobilizations. Massage therapy. Suboccipital inhibition. Once a week.
  Interventions: Other: Physical Therapy
- Therapeutic Exercise Group (Experimental): Recruitment and strengthening of the cervical flexors. Isometric cervical exercises with self-resistance. Shoulder girdle strengthening exercise. Alternating days.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — A manual therapy protocol and a therapeutic exercise protocol

SUMMARY:
It has been estimated that between 50% and 85% of the population will suffer neck pain along their life. Chronic nonspecific neck pain is one of the main causes of disability in the population, it represents 25% of visits to physiotherapy, and it also has a high chance of chronification. The efficacy of combining manual therapy and therapeutic exercise for the treatment of this pathology has been demonstrated a lot of times. However, no conclusive studies have been found that compare the isolated application of both treatments, thus being an important focus of action and research.

The main objective of the study is to check if the treatment with therapeutic exercise is better than manual therapy in the improvement of the disability in patients with chronic neck pain.

A randomized, controlled, monocentric, parallel and single-blind clinical trial will be carried out.

The simple will be obtained from the population over 18 years old with chronic neck pain of more than 12 weeks of evolution and will be those who meet the inclusion and exclusion criteria.

The patients will be randomly divided into 2 intervention groups, in one of the groups will be applied a manual therapy session of about 30 minutes once a week for 4 weeks. In the other group it will be delivered and explained to the patients, a home therapeutic exercise program that will be carried out on alternate days for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific cervical pain of more than 12 weeks of evolution.
* Over 18 years.

Exclusion Criteria:

* Oncological processes.
* Pregnancy.
* Infectious diseases.
* Degenerative diseases.
* Fibromyalgia.
* Previous spinal surgeries.
* Previous traumatic events.
* Hernias and/or cervical protrusions.
* Neurological processes.
* Current treatment for cervical pain.
* Neuropathic characteristics pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | Three months

SECONDARY OUTCOMES:
Visual Analog Scale | Three months
Pressure Pain Threshold | Three months
Life Quality SF-12 | Three months
Kinesiophobia TAMPA Scale | Three months
Beck Depression Inventory II | Three months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alcala, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No